CLINICAL TRIAL: NCT00922701
Title: Phase 2 Study of Dialysis Efficiency and Tolerability of Nocturnal Peritoneal Dialysis Solution Containing Glucose Plus L-carnitine
Brief Title: L-Carnitine in Peritoneal Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Arduino Arduini, MD, Iperboreal Pharma Srl
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-001-04
Record Dates: First submitted 2009-02-11; First posted 2009-06-17 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: End-Stage Renal Disease
Keywords: Peritoneal dialysis; L-carnitine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peritoneal Dialysis Solution (Experimental)
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — Instillation of glucose-based (1.5% weight/volume) peritoneal dialysis solution containing L-carnitine (0.25% weight/volume) for the nocturnal exchange. Patients were treated with the experimental peritoneal dialysis solution for 5 days.

SUMMARY:
The development of glucose-sparing strategies able to provide an efficacious ultrafiltration profile represents one of the modern goals of peritoneal dialysis therapy. The study hypothesis is to evaluate the possibility to formulate peritoneal dialysis solutions containing L-carnitine as an osmotic agent to partially replace glucose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Have a diagnosis of End Stage Renal Disease and have been on Continuous Ambulatory Peritoneal Dialysis for at least 3 months
* Be in a stable clinical condition during the four weeks immediately prior to Screening Period as demonstrated by medical history, physical examination and laboratory testing
* Have a blood hemoglobin concentration above 8,5 g/100ml (data will be verified with Investigators)
* Have not experienced peritonitis episodes in the last 3 months
* Be treated with 3 diurnal exchange bag solutions (1.5% or 2.5% glucose) and one nocturnal exchange bag solution (2.5% glucose)
* Have Kt/V urea measurement > 1.7 per week in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a minimum weekly creatinine clearance of 45 litres in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a D/P Creatinine ratio at Peritoneal Equilibration Test between 0.50 and 0.81 in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a D/P Glucose ratio at Peritoneal Equilibration Test between 0.26 and 0.49 in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Be treated by the participating clinical Investigator for a period of at least three months
* Have understood and signed the Informed Consent Form.

Exclusion Criteria:

* Have a history of drug or alcohol abuse in the six months prior to entering the protocol
* Be in treatment with androgens
* Have Diabetes Mellitus (as defined by the American Diabetes Society, objectively documented by a fasting plasma glucose and HbA1c determinations)
* Have clinically significant abnormal liver function test (SGOT, SGPT, and gamma-GT > 2 times the upper normal limit)
* Have acute infectious conditions (i.e.: pulmonary infection, acute hepatitis, high or low urinary tract infections, renal parenchymal infection, pericarditis, etc)
* Have a history of congestive heart failure and clinically significant arrhythmia
* Have an history of epilepsy or any central nervous system disease
* Have malignancy within the past 5 years, including lymphoproliferative disorders
* Have any medical condition that, in the judgment of the Investigator, would jeopardize the patient's safety following exposure to study drug, particularly if patient's life expectancy is less than 1 year
* Have a history of L-Carnitine therapy or use in the month prior to entering the protocol
* Have used any investigational drug in the 3 months prior to entering the protocol
* Pregnant, lactating, fertility age without protection against pregnancy by adequate contraceptive means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-06; Primary Completion 2004-10 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bonomini, M.D., Principal Investigator — G. d'Annunzio University; Arduino Arduini, M.D., Study Director — Iperboreal Pharma Srl
Locations (1):
- Division of Nephrology, University of "G. d'Annunzio", Chieti, Italy

REFERENCES:
- [Derived] Bonomini M, Pandolfi A, Di Liberato L, Di Silvestre S, Cnops Y, Di Tomo P, D'Arezzo M, Monaco MP, Giardinelli A, Di Pietro N, Devuyst O, Arduini A. L-carnitine is an osmotic agent suitable for peritoneal dialysis. Kidney Int. 2011 Sep;80(6):645-54. doi: 10.1038/ki.2011.117. Epub 2011 Apr 27. PMID 21525850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June, 2004, to November, 2004. Medical Clinic
Pre-assignment Details: One-week run-in
Groups:
- Peritoneal Dialysis Solution: Patients were treated with a glucose-based (1.5% weight/volume) peritoneal dialysis solution containing L-carnitine (0.25% weight/volume) for the long dwell. Peritoneal dialysis solution was instilled for 5 days.
Period: Overall Study
Arm/Group | Peritoneal Dialysis Solution
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Peritoneal Dialysis Solution: The enrolled patients were using for the long dwell (nocturnal) exchange a glucose-based (2.5% w/v) peritoneal dialysis solution.
Arm/Group | Peritoneal Dialysis Solution
Number analyzed (Participants) | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  Italy | 4
Ultrafiltration [Mean (Standard Deviation); unit: milliliters] — Ultrafiltration measured at the end of the long dwell (nocturnal) exchange
  milliliters | 1987 (192)

OUTCOME MEASURES:

1. Primary Outcome: Long Dwell Ultrafiltration
Description: The amount of fluid recovered from the peritoneum at the end of the nocturnal exchange (long dwell) with a peritoneal dialysis solution.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Peritoneal Dialysis Solution
Number analyzed (Participants) | 4
milliliters | 2167 (203)

ADVERSE EVENTS:
Arm/Group | Peritoneal Dialysis Solution
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No